CLINICAL TRIAL: NCT00712426
Title: Creatine Safety, Tolerability, & Efficacy in Huntington's Disease (CREST-E)
Acronym: CREST-E
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Results of an interim analysis showed that it was unlikely that creatine was effective in slowing loss of function in early symptomatic Huntington's Disease.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Rochester (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Steven M. Hersch, Professor of Neurology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007P000827; U01AT000613 (NIH)
Record Dates: First submitted 2008-07-08; First posted 2008-07-10 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-02

CONDITIONS: Huntington's Disease
Keywords: Huntington's disease; Creatine; Mitochondrial Dysfunction; Total Functional Capacity; UHDRS
MeSH Terms: conditions — Huntington Disease; Mitochondrial Diseases | interventions — Creatine; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Randomized to receive creatine monohydrate (up to 40 grams daily)
  Interventions: Drug: Creatine Monohydrate
- B (Placebo Comparator): Randomized to receive placebo (up to 40 grams daily)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Creatine Monohydrate — Up to 40 grams daily, powder form creatine monohydrate, taken for the trial duration
  Other Names: HD-02
  Arms: A
Drug: Placebo — Up to 40 grams daily, powder form placebo (inactive substance), taken for the trial duration
  Other Names: Dextrose
  Arms: B

SUMMARY:
Huntington's disease (HD) is a slowly progressive disorder that devastates the lives of those affected and their families. There are no treatments that slow the progression of HD, only mildly effective symptomatic therapies are available.Creatine monohydrate is considered a nutritional supplement. The purpose of CREST-E is to test whether high-dose creatine can slow the progressive functional decline that occurs in persons 18 years or older with early clinical features of HD. The long-term safety, tolerability and effectiveness of up to 40 grams daily creatine compared to placebo is studied. A variety of biological processes are assessed for markers of disease activity or progression and creatine effects. Up to 50 active research centers globally will enroll 650 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ages 18 or older.
* Clinical features of HD AND confirmatory family history of HD; OR Clinical features of HD AND CAG repeat expansion greater or equal to 36.
* Stage I or II of illness (TFC greater or equal to 7).
* Ambulatory and not requiring skilled nursing care at the time of enrollment.
* Must be capable of providing informed consent and complying with trial procedures.
* Additional inclusion criteria apply.

Exclusion Criteria:

* History of known sensitivity or intolerability to creatine monohydrate.
* Exposure to any investigational drug within 30 days of randomization (Baseline visit).
* Use of supplemental creatine at a dose greater than 10 grams within 30 days of randomization (Baseline visit).
* Screening laboratory abnormalities that in the judgment of the investigator would jeopardize safe conduct of study.
* Clinical evidence of unstable medical illness.
* Clinical evidence of unstable psychiatric illness.
* Additional exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 553 (Actual)
Dates: Start 2009-09; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in Total Functional Capacity | Minimum 12 months up to 48 months
  Study duration depends on each subject's calendar date of enrollment.

SECONDARY OUTCOMES:
Clinical symptoms (changes in other UHDRS scores); safety (frequency of adverse events); tolerability (proportion of subjects completing study at assigned dosage level), quality of life, other biological markers. | Duration of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Hersch, MD, PhD, Principal Investigator — Massachusetts General Hospital; Giovanni Schifitto, MD, Principal Investigator — University of Rochester Clinical Trial Coordination Center; Diana Rosas, MD, MS, Principal Investigator — Massachusetts General Hospital
Locations (47):
- United States (38):
  - University of Alabama, Birmingham, Alabama
  - University of California, Irvine, Irvine, California
  - University of California Davis, Sacramento, California
  - University of Connecticut, Farmington, Connecticut
  - University of Florida (McKnight Brain Institute), Gainesville, Florida
  - University of South Florida, Tampa, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Georgia Regents University, Augusta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Hereditary Neurological Disease Center (HNDC), Wichita, Kansas
  - University of Louisville, Louisville, Kentucky
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Struthers Parkinson's Center, Golden Valley, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Medical Center, Omaha, Nebraska
  - Cooper University Hospital, Camden, New Jersey
  - Albany Medical College, Albany, New York
  - North Shore-LIJ Health System, Manhasset, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Duke University, Durham, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Booth Gardner Parkinson's Care Center (Evergreen Healthcare), Kirkland, Washington
- Australia (2):
  - Westmead Hospital, Wentworthville, New South Wales
  - Neurodegenerative Disorders Research, Subiaco, Western Australia
- Canada (5):
  - University of Alberta Hospital, Edmonton, Alberta
  - University of Alberta, Edmonton, Alberta
  - Movement Disorder Clinic Deer Lodge Center, Winnipeg, Manitoba
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - University of Quebec Infant-Jesus Hospital (Centre Hospitalier Affilie), Québec, Quebec
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - New Zealand Brain Research Institute, Christchurch

REFERENCES:
- [Background] Kim J, Amante DJ, Moody JP, Edgerly CK, Bordiuk OL, Smith K, Matson SA, Matson WR, Scherzer CR, Rosas HD, Hersch SM, Ferrante RJ. Reduced creatine kinase as a central and peripheral biomarker in Huntington's disease. Biochim Biophys Acta. 2010 Jul-Aug;1802(7-8):673-81. doi: 10.1016/j.bbadis.2010.05.001. Epub 2010 May 9. PMID 20460152
- [Background] Hersch SM, Gevorkian S, Marder K, Moskowitz C, Feigin A, Cox M, Como P, Zimmerman C, Lin M, Zhang L, Ulug AM, Beal MF, Matson W, Bogdanov M, Ebbel E, Zaleta A, Kaneko Y, Jenkins B, Hevelone N, Zhang H, Yu H, Schoenfeld D, Ferrante R, Rosas HD. Creatine in Huntington disease is safe, tolerable, bioavailable in brain and reduces serum 8OH2'dG. Neurology. 2006 Jan 24;66(2):250-2. doi: 10.1212/01.wnl.0000194318.74946.b6. PMID 16434666
- [Background] Ryu H, Rosas HD, Hersch SM, Ferrante RJ. The therapeutic role of creatine in Huntington's disease. Pharmacol Ther. 2005 Nov;108(2):193-207. doi: 10.1016/j.pharmthera.2005.04.008. Epub 2005 Aug 1. PMID 16055197
- [Background] Dedeoglu A, Kubilus JK, Yang L, Ferrante KL, Hersch SM, Beal MF, Ferrante RJ. Creatine therapy provides neuroprotection after onset of clinical symptoms in Huntington's disease transgenic mice. J Neurochem. 2003 Jun;85(6):1359-67. doi: 10.1046/j.1471-4159.2003.01706.x. PMID 12787055
- [Background] Andreassen OA, Dedeoglu A, Ferrante RJ, Jenkins BG, Ferrante KL, Thomas M, Friedlich A, Browne SE, Schilling G, Borchelt DR, Hersch SM, Ross CA, Beal MF. Creatine increase survival and delays motor symptoms in a transgenic animal model of Huntington's disease. Neurobiol Dis. 2001 Jun;8(3):479-91. doi: 10.1006/nbdi.2001.0406. PMID 11447996
- [Background] Ferrante RJ, Andreassen OA, Jenkins BG, Dedeoglu A, Kuemmerle S, Kubilus JK, Kaddurah-Daouk R, Hersch SM, Beal MF. Neuroprotective effects of creatine in a transgenic mouse model of Huntington's disease. J Neurosci. 2000 Jun 15;20(12):4389-97. doi: 10.1523/JNEUROSCI.20-12-04389.2000. PMID 10844007
- [Derived] McGarry A, Auinger P, Kieburtz KD, Bredlau AL, Hersch SM, Rosas HD. Suicidality Risk Factors Across the CARE-HD, 2CARE, and CREST-E Clinical Trials in Huntington Disease. Neurol Clin Pract. 2022 Apr;12(2):131-138. doi: 10.1212/CPJ.0000000000001161. PMID 35747889
- [Derived] Rodrigues FB, Wild EJ. Huntington's Disease Clinical Trials Corner: August 2018. J Huntingtons Dis. 2018;7(3):279-286. doi: 10.3233/JHD-189003. PMID 30103342
- [Derived] Hersch SM, Schifitto G, Oakes D, Bredlau AL, Meyers CM, Nahin R, Rosas HD; Huntington Study Group CREST-E Investigators and Coordinators. The CREST-E study of creatine for Huntington disease: A randomized controlled trial. Neurology. 2017 Aug 8;89(6):594-601. doi: 10.1212/WNL.0000000000004209. Epub 2017 Jul 12. PMID 28701493
- See also: Huntington Study Group (CREST-E Study) — http://www.huntington-study-group.org/ClinicalResearch/ClinicalTrialsObservationalStudiesinProgress/CRESTE/tabid/105/Default.aspx